CLINICAL TRIAL: NCT06944587
Title: A New Clinical Pathway for Personalized Management of Borderline Resectable and Locally Advanced Pancreatic Cancer - Norwegian Pancreatic Cancer Trial-3 (NORPACT 3)
Brief Title: A New Clinical Pathway for Personalized Management of Borderline Resectable and Locally Advanced Pancreatic Cancer
Acronym: NORPACT-3
Status: Recruiting | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: University Hospital of North Norway (Other); Haukeland University Hospital (Other); Helse Stavanger HF (Other Government); St.Olavs Hospital, Trondheim University Hospital, Norway (Unknown)
Responsible Party: Principal Investigator, Knut Jørgen Labori, Professor of Surgery, Senior consultant surgeon, Oslo University Hospital
Other Study IDs: REK sør-øst D 733339; 2023010 (Other Grant/Funding Number: Southern and Eastern Norway Regional Health Authority); 279530-2023 (Other Grant/Funding Number: Norwegian Cancer Society)
Record Dates: First submitted 2025-01-17; First posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Locally Advanced Pancreatic Cancer; Borderline Resectable Pancreatic Cancer; Pancreatectomy; Chemotherapy Effect
Keywords: Primary chemotherapy; Resection rate; Borderline Resectable Pancreatic Cancer; Locally Advanced Pancreatic Cancer; Pancreatectomy; Chemotherapy Effect; FDG PET-CT; ctDNA
MeSH Terms: interventions — Drug Therapy; Diagnostic Imaging; Tomography, X-Ray Computed; Pancreatectomy; Endoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples for circulating tumor DNA analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Chemotherapy — The choice of chemotherapy regimen follows national guidelines, preferably mFOLFIRINOX or gemcitabine-nab-paclitaxel.
Diagnostic Test: Radiology — PET/CT is optional. PET/CT will be offered as a part of the diagnostic work up at baseline and one additional scan after a minimum of two months of chemotherapy.
  Other Names: Fluorine-18-fluorodeoxyglucose positron emission/computed tomography
Procedure: Pancreatectomy — Surgery is scheduled within 4 weeks after the last neoadjuvant infusion. Resection will be performed as a standard or pylorus-preserving pancreatoduodenectomy (PD), distal pancreatectomy (DP) with splenectomy, or total pancreatectomy (TP) with splenectomy, and with or without venous or arterial resection and reconstruction.
Procedure: Endoscopy — Endoscopic ultrasound fine-needle biopsy to establish the diagnosis with histopathology and to obtain an adequate sample for molecular pathology (KRAS status (mutation or wild type), microsatellite instability (MSI)).

SUMMARY:
NORPACT-3 is a nationwide, Norwegian single arm prospective study that evaluates the resectability rates and survival in patients with borderline resectable and locally advanced pancreatic cancer who received primary chemotherapy. Eligible patients are treated with primary chemotherapy possibly followed by surgical exploration and resection. All Norwegian centres performing pancreatic surgery have agreed to collaborate in this trial. The assignment of the medical intervention is not at the discretion of the investigator, but follow the national Norwegian guidelines regarding diagnostic work up, oncological and surgical treatment and follow up. The primary aim is a national resection rate of 50% in BRPC and 15% in LAPC in patients initiating primary chemotherapy, with adequate overall survival and morbidity/mortality (after resection median overall survival of 24 months, 1 year survival 80%, and 5 year survival >20% + 90 day postoperative mortality ≤5%, 90-day postoperative major morbidity (Clavien Dindo grade 3) ≤40%).

ELIGIBILITY:
Inclusion Criteria:

* Borderline resectable or locally advanced adenocarcinoma of the pancreas (NCCN, version 2, 2021) (Appendix 3)
* Nx, M0 (UICC 8th version, 2016)
* Cytological or histological confirmation of adenocarcinoma
* Age >18 year
* Considered able to receive primary chemotherapy and possible surgery
* Written informed consent

Exclusion Criteria:

* Co-morbidity or performance status precluding primary chemotherapy
* Co-morbidity or performance status precluding pancreatectomy
* Female patients in child-bearing age not using adequate contraception, pregnant or lactating women
* Mental or physical disorders that could interfere with treatment of with the provision of informed consent
* Any reason why, in the opinion of the investigator, the patient should not participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Nationwide, population based cohort from a universal health care system
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-12-03 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Resection rate (of the pancreatic tumour) | From November 2024-December 2027
  Resection rate: National target of 50% in BRPC and 15% in LAPC in patients initiating primary chemotherapy.

SECONDARY OUTCOMES:
Overall survival | From November 2024-December 2027
  After resection, median overall survival of 24 months, 1 year survival 80%, and 5 year survival >20%.
Mortality after surgical resection | From November 2024-December 2027
  90-day postoperative mortality ≤5%
Morbidity after surgical resection | From November 2024-December 2027
  90-day postoperative major morbidity (Clavien-Dindo ≥ grade3) of ≤40%
Number of patients evaluated at national MDT undergoing resection | From November 2024-December 2027
Adverse events | From November 2023-December 2027
  Adverse events during primary chemotherapy
R0 resection rate | From November 2023-December 2027
  R0 (microscopic radical resection >1mm) versus R1 (microscopic residual tumor ≤1mm).
Quality of life EORTC QLQ-C30 | Measured at baseline, 3, 6, and 12 months from diagnosis, followed by yearly measurements.]
  Outcome measures will be calculated, according to the validated questionnaire manuals.
Quality of life EORTC QLQ-PAN26 | Measured at baseline, 3, 6, and 12 months from diagnosis, followed by yearly measurements.
  Outcome measures will be calculated, according to the validated questionnaire manuals.
Quality of life EQ-5D-5L | Measured at baseline, 3, 6, and 12 months from diagnosis, followed by yearly measurements.
  Outcome measures will be calculated, according to the validated questionnaire manuals.

OTHER OUTCOMES:
PET CT | From November 2023-December 2027
  * Extrapancreatic disease detected at baseline PET-CT
  * Correlation of PET-CT findings with histopathological tumor regression grading
  * Correlation of PET-CT findings with CA19-9 dynamics
  * Prognostic value of metabolic tumor response in resected patients
Molecular profiling (KRAS mutation status, MSI) at time of diagnosis | From November 2023-December 2027
  * Number of patients with KRAS mutations, KRAS wild type, or MSI tumors
  * Number of patients undergoing additional genetic profiling and/or targeted therapy in accordance with the national guidelines protocols or ongoing trials.

CONTACTS AND LOCATIONS:
Locations (5):
- Norway (5):
  - Haukeland University Hospital, Bergen, Norway
  - Stavanger University Hospital, Stavanger, Norway
  - University Hospital of North Norway, Tromsø, Norway
  - St. Olavs Hospital, Trondheim University Hospital, Trondheim, Norway
  - Oslo University Hospital, Oslo

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Boggi U, Kauffmann EF, Napoli N, Barreto SG, Besselink MG, Fusai GK, Hackert T, Hilal MA, Marchegiani G, Salvia R, Shrikhande SV, Truty M, Werner J, Wolfgang C, Bannone E, Capretti G, Cattelani A, Coppola A, Cucchetti A, De Sio D, Di Dato A, Di Meo G, Fiorillo C, Gianfaldoni C, Ginesini M, Hidalgo Salinas C, Lai Q, Miccoli M, Montorsi R, Pagnanelli M, Poli A, Ricci C, Sucameli F, Tamburrino D, Viti V, Cameron J, Clavien PA, Asbun HJ; REDISCOVER guidelines group. REDISCOVER guidelines for borderline-resectable and locally advanced pancreatic cancer: management algorithm, unanswered questions, and future perspectives. Updates Surg. 2024 Sep;76(5):1573-1591. doi: 10.1007/s13304-024-01860-0. Epub 2024 Apr 29. PMID 38684573
- [Background] Springfeld C, Ferrone CR, Katz MHG, Philip PA, Hong TS, Hackert T, Buchler MW, Neoptolemos J. Neoadjuvant therapy for pancreatic cancer. Nat Rev Clin Oncol. 2023 May;20(5):318-337. doi: 10.1038/s41571-023-00746-1. Epub 2023 Mar 17. PMID 36932224
- [Background] Stoop TF, Theijse RT, Seelen LWF, Groot Koerkamp B, van Eijck CHJ, Wolfgang CL, van Tienhoven G, van Santvoort HC, Molenaar IQ, Wilmink JW, Del Chiaro M, Katz MHG, Hackert T, Besselink MG; International Collaborative Group on Locally Advanced Pancreatic Cancer. Preoperative chemotherapy, radiotherapy and surgical decision-making in patients with borderline resectable and locally advanced pancreatic cancer. Nat Rev Gastroenterol Hepatol. 2024 Feb;21(2):101-124. doi: 10.1038/s41575-023-00856-2. Epub 2023 Nov 30. PMID 38036745
- [Background] Farnes I, Kleive D, Verbeke CS, Aabakken L, Issa-Epe A, Smastuen MC, Fosby BV, Dueland S, Line PD, Labori KJ. Resection rates and intention-to-treat outcomes in borderline and locally advanced pancreatic cancer: real-world data from a population-based, prospective cohort study (NORPACT-2). BJS Open. 2023 Nov 1;7(6):zrad137. doi: 10.1093/bjsopen/zrad137. PMID 38155512